CLINICAL TRIAL: NCT02567565
Title: Evaluation of Tear Film Lipid Layer Thickness Change After Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0225
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Cataract Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cataract patients: cataract patients undergoing phacoemulsification
  Interventions: Other: LipiView

INTERVENTIONS:
Other: LipiView — tear film lipid layer thickness measured by LipiView interferometer (TearScience Inc, Morrisville, NC)

SUMMARY:
This study will compare cataract patients before and after phacoemulsification. Evaluations will be performed before and 1 and 3 months following cataract surgery, including measurement of tear film lipid layer thickness, tear film break up time, Schirmer test, corneal and conjunctival fluorescein staining, examination of lid margins and meibomian glands, and the Ocular Surface Disease Index.

ELIGIBILITY:
Inclusion Criteria:

* cataract patients with lens opacities classification higher than grade III and desire to be spectacle independence for distance and near vision

Exclusion Criteria:

* previous ocular surgery or trauma and the presence of corneal opacities, fundus abnormalities, glaucoma, uveitis, amblyopia, systemic disease, and posterior capsule rupture during cataract surgery

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cataract patients with lens opacities classification higher than grade III
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
tear film lipid layer thickness | 3-month after phacoemulsification
  tear film lipid layer thickness measured by LipiView interferometer

CONTACTS AND LOCATIONS:
Overall Officials: Tae-im Kim, MD, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Department of Ophthalmology, Yonsei University College of Medicine, Seoul, Seoul, South Korea